CLINICAL TRIAL: NCT07381179
Title: Voices: Messages of Wisdom and Hope in the Face of Illness
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 25-006417; NCI-2026-00073 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-006417 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2026-01-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients and their caregivers complete an interview and survey on study. Patients also have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study may help doctors determine where patients and caregivers may need more support and identify ways to maintain patient and caregiver dignity while undergoing treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Change in patient dignity impact scale scores prior to and after completion of patient and caregiver recordings.

OUTLINE: This is an observational study.

Patients and their caregivers complete an interview and survey on study. Patients also have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of chronic or progressive illness with a primary caregiver, should patient wish to involve one
* Willing and able to participate in a semi-structured recording lasting approximately 60 minutes. Dyad recordings conducted for participants who elect to involve a caregiver
* Willing and able to participate in a single follow-up recording. Dyad follow up recordings conducted for participants who elect to involve a caregiver

Exclusion Criteria:

* Uncontrolled and/or intercurrent illness which limits participation in study recording
* Vulnerable populations: persons lacking capacity for understanding participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosis of chronic or progressive illness with a primary caregiver, should patient wish to involve one.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-12-13 (Estimated); Study Completion 2027-12-13 (Estimated)

PRIMARY OUTCOMES:
Change in patient dignity impact | Baseline (before and after recording)
  Will assess patient dignity impact scale scores prior to and after completion of patient and caregiver recordings. The dignity impact scale (DIS) is a 7-item questionnaire with responses scaling from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate greater levels of dignity. Patient participants will complete the survey before and after their recordings as outlined in the schedule of events. Surveys will be completed digitally.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur Sener, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials